CLINICAL TRIAL: NCT00073411
Title: Duloxetine Versus Escitalopram and Placebo in the Treatment of Patients With Major Depression
Brief Title: Duloxetine Compared to Escitalopram and Placebo in the Treatment of Patients With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7978; F1J-US-HMCR
Record Dates: First submitted 2003-11-20; First posted 2003-11-21 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: duloxetine
Drug: escitalopram
Drug: placebo

SUMMARY:
The purposes of this study are to determine:

* The safety of duloxetine and any side effects that might be associated with it.
* How duloxetine compares to escitalopram and placebo (an inactive ingredient)

DETAILED DESCRIPTION:
duloxetine 60mg - 120mg, escitalopram 10mg - 20mg, and placebo, 8-month,

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 of age
* Must meet the criteria for major depressive disorder
* You must be able to visit the doctor's office about once a week for 2 to 3 months. After that, you will need to visit the doctor's office once a month for about 6 months
* You must be able to take the study drug as prescribed (6 capsules per day taken once-daily)

Exclusion Criteria:

* You are a woman and are pregnant or breastfeeding.
* You have a current or previous major psychiatric disorder other than depression, such as bipolar disorder, schizophrenia, or other psychotic disorder.
* You have a history of alcohol or drug dependence within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675
Dates: Start 2003-11; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To compare the onset of antidepressant efficacy for duloxetine 60 mg once-daily compared with escitalopram 10 mg once-daily.

SECONDARY OUTCOMES:
To compare the efficacy of duloxetine 60 mg once-daily versus escitalopram 10 mg once-daily and placebo during acute therapy
To compare the efficacy of duloxetine 60-120 mg once-daily versus escitalopram 10-20 mg once-daily and placebo for up to 8 months of therapy
To compare incidence of sexual dysfunction (defined by Changes in Sexual Functioning Questionnaire (CSFQ)), during acute therapy for patients treated with duloxetine 60 mg once-daily versus escitalopram 10 mg once-daily & placebo.
To compare sexual dysfunction during up to 8 months of treatment with duloxetine 60-120 mg once-daily versus escitalopram 10 to 20 mg once-daily and placebo
To compare impact of duloxetine 60 mg once-daily versus escitalopram 10 mg once-daily & placebo during acute therapy & during 8 months of therapy on quality of life, functional/health outcomes, & patient satisfaction with study drug
To compare impact of duloxetine 60-120 mg once-daily versus escitalopram 10 to 20 mg once-daily and placebo for up to 8 months of therapy on quality of life, functional/health outcomes, & patient satisfaction with study drug
To compare impact of duloxetine 60-120 mg once-daily versus escitalopram 10-20 mg once-daily and placebo during acute and extended therapy on resource utilization (% patients using more,less or equal number of health care providers and services)
To evaluate safety and tolerability of duloxetine 60 mg once-daily vs. escitalopram 10 mg once-daily and placebo during acute therapy
To evaluate the safety and tolerability of duloxetine 60-120 mg once-daily vs. escitalopram 10-20 mg once-daily and placebo for up to 8 months of therapy
To compare percentage of patients taking duloxetine 60 mg once-daily versus escitalopram 10 mg once-daily and placebo requiring a dose escalation due to less than satisfactory initial response (defined by IRB supplement or investigator request)
To compare efficacy of duloxetine versus escitalopram in the placebo non-responders who enter the rescue phase

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Harada E, Kato M, Fujikoshi S, Wohlreich MM, Berggren L, Tokuoka H. Changes in energy during treatment of depression: an analysis of duloxetine in double-blind placebo-controlled trials. Int J Clin Pract. 2015 Oct;69(10):1139-48. doi: 10.1111/ijcp.12658. Epub 2015 May 16. PMID 25980552
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392
- [Derived] Gueorguieva R, Mallinckrodt C, Krystal JH. Trajectories of depression severity in clinical trials of duloxetine: insights into antidepressant and placebo responses. Arch Gen Psychiatry. 2011 Dec;68(12):1227-37. doi: 10.1001/archgenpsychiatry.2011.132. PMID 22147842
- [Derived] Sheehan DV, Harnett-Sheehan K, Spann ME, Thompson HF, Prakash A. Assessing remission in major depressive disorder and generalized anxiety disorder clinical trials with the discan metric of the Sheehan disability scale. Int Clin Psychopharmacol. 2011 Mar;26(2):75-83. doi: 10.1097/YIC.0b013e328341bb5f. PMID 21102344
- [Derived] Prakash A, Risser RC, Mallinckrodt CH. The impact of analytic method on interpretation of outcomes in longitudinal clinical trials. Int J Clin Pract. 2008 Aug;62(8):1147-58. doi: 10.1111/j.1742-1241.2008.01808.x. Epub 2008 Jun 28. PMID 18564199
- [Derived] Pigott TA, Prakash A, Arnold LM, Aaronson ST, Mallinckrodt CH, Wohlreich MM. Duloxetine versus escitalopram and placebo: an 8-month, double-blind trial in patients with major depressive disorder. Curr Med Res Opin. 2007 Jun;23(6):1303-18. doi: 10.1185/030079907X188107. Epub 2007 Apr 27. PMID 17559729
- [Derived] Nierenberg AA, Greist JH, Mallinckrodt CH, Prakash A, Sambunaris A, Tollefson GD, Wohlreich MM. Duloxetine versus escitalopram and placebo in the treatment of patients with major depressive disorder: onset of antidepressant action, a non-inferiority study. Curr Med Res Opin. 2007 Feb;23(2):401-16. doi: 10.1185/030079906X167453. PMID 17288694
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com